CLINICAL TRIAL: NCT02758704
Title: Impact of Stress on the Performance of Neonatal Endotracheal Intubation: A Randomized Controlled Trial on Manikins
Brief Title: Impact of Stress on Performance of Neonatal Endotracheal Intubation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Justine's Hospital (Other)
Collaborators: Alberta Children's Hospital (Other)
Responsible Party: Principal Investigator, Ahmed Moussa, Neonatologist, Clinical assistant professor, St. Justine's Hospital
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: 4143
Record Dates: First submitted 2016-04-27; First posted 2016-05-02 (Estimated); Last update posted 2021-10-07 (Actual); Status verified 2021-10

CONDITIONS: Neonatal Intubation Performance
Keywords: Intubation; Neonatal; Teaching; Stress; Simulation
MeSH Terms: interventions — RCF3 protein, Arabidopsis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- High-Stress (HS) (Experimental): In the HS environment, the resident will be exposed to various stressors. There will be the presence of audio alarms as well as the presence of a senior physician who will be supervising the performance of the resident. In addition, the mannequin will be slightly unstable which will be reflected in its oxygen saturation dropping throughout the first 30 seconds the procedure.
  Interventions: Other: High stress; Other: Endotracheal intubation on mannequin
- Low-Stress (LS) (Active Comparator): In the LS environment, there will be absence of audio (alarms), physical (third-party supervisor, nurse and respiratory therapist) and situational (unstable infant) stressors.
  Interventions: Other: Low stress; Other: Endotracheal intubation on mannequin

INTERVENTIONS:
Other: High stress — Generation of a stressful environment during a neonatal intubation procedure.
  Arms: High-Stress (HS)
Other: Low stress — Absence of stressful stimuli during neonatal intubation procedure
  Arms: Low-Stress (LS)
Other: Endotracheal intubation on mannequin — Endotracheal intubation will take place at the simulation centre on a mannequin.

SUMMARY:
This study will be a randomized controlled trial designed to analyse the impact of stress on the success rate of a simulated neonatal endotracheal intubation. To do this, pediatric residents will be enrolled and randomized to either a high-stress (HS) or low-stress (LS) environment where they will be asked to perform a standard neonatal intubation procedure. Subjects will then cross-over to the second scenario within a short window (1-2 weeks). Outcome measures include: endotracheal intubation success rate and assessment of the procedure performance by video-review using a standardized checklist rated by two independent reviewers. Stress level will be measured using salivary cortisol, heart rate and a standardized anxiety questionnaire.

DETAILED DESCRIPTION:
Although a required skill in pediatric residency programs, success rate of neonatal endotracheal intubation (ETI) among trainees is known to be inadequate. Currently, it is taught using simulation; a teaching method that seems useful mainly for limited short-term retention of skill. In the clinical setting, ETI is often associated with stress, which could explain the limited educational impact of simulation training. The effect of stress on the success of this procedure is poorly studied.

Therefore, the objective of the investigators study is to assess the impact of stress on the success of simulated neonatal ETI.

Hypotheses to be tested: The primary hypothesis is that stressful conditions will negatively impact residents' success of endotracheal intubation on neonatal manikins. Secondary hypotheses include: 1) stressful conditions will be associated with an increased time to successful intubation and decreased performance on the intubation checklist; 2) there will be a positive correlation between heart rate/cortisol levels and resident's response on the State Trait Anxiety Inventory questionnaire (STAI).

Design: This study will be a crossover randomized controlled trial in the setting of the simulation laboratory. Subjects will include pediatric residents and pediatric subspecialty residents. Exclusion criteria will include any medical condition or medication that can have a significant impact on cortisol levels. The residents will be randomized using sealed envelopes to perform a neonatal ETI in a low or a high stress environment, and then crossover to the other on a separate day. Stress will be created and standardized by using audio alarms, third party supervisors and simulated manikin instability. Level of stress of participants will be assessed at baseline during a lecture, upon arrival to the simulation center and after the simulated procedure. This will be done using salivary cortisol, heart rate and the STAI questionnaire. ETI procedures will be videotaped and performance will be assessed by two external reviewers using a validated checklist.

Analysis: Primary and secondary outcomes include: success rate, checklist performance, time to successful intubation, rate of esophageal intubation and stress levels (cortisol, heart rate and questionnaire). Continuous variables will be analyzed by the independent sample t test and categorical variables will be analyzed by Fisher's exact test. Statistical significance will be defined by a 2-sided alpha of 0.05 and power of 80%. To demonstrate a decrease of success rate of ETI from 80% (retrieved from previous simulation study in a LS environment) to 60%, 64 intubations are needed per group.

Anticipated outcomes & potential problems: Demonstrating a decrease in success rate of ETI in the HS environment will aid to improve simulation-based training of neonatal ETI. In the future, the HS environment model can be used as an intermediate training process to prepare residents to the stress related to this procedure in the clinical world.

ELIGIBILITY:
Inclusion Criteria:

* All residents enrolled in the pediatric residency program and subspecialties of University of Montreal.

Exclusion Criteria:

* Residents who have a medical condition that can impact cortisol levels, such as pregnancy, will be excluded from the cortisol analysis.

Max Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 58 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Success rate of endotracheal intubation procedure | 5 minutes
  Successful intubation will be defined as correct placement of the endotracheal tube just below the level of the vocal cords and will be verified by one of the investigators at the end of the procedure. Each attempt will be limited to 30 sec, as per Neonatal Resuscitation Program guidelines. An esophageal intubation will be defined as the absence of chest rise upon completion of the procedure.
Intubation skill performance | within 24 months
  Endotracheal intubation procedures will be videotaped and performance will be assessed by two external reviewers using an ETI checklist (in the process of validation).

SECONDARY OUTCOMES:
Rate of esophageal intubation | 5 minutes
Stress level - Cortisol Measurement | within 24 months
  At rest, before and after each scenario
Stress level - Heart Rate | within 24 months
  At rest, before and after each scenario
Stress level - STAI Questionnaire | within 24 months
  Subjects will be asked to fill out the State-Trait Anxiety Inventory questionnaire at rest, prior to and after each simulation scenario
Duration of intubation | 5 minutes
  Timing will begin when the laryngoscope's blade is inserted into the manikin's mouth. The end of the attempt is indicated by the laryngoscope blade leaving the mannikin's mouth.

CONTACTS AND LOCATIONS:
Locations (2):
- Canada (2):
  - Alberta Children's Hospital, Calgary, Alberta
  - Sainte-Justine Hospital, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: Yes